CLINICAL TRIAL: NCT05942482
Title: Head and Neck Paragangliomas: A 16-year Experience of a University Hospital in Turkey
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Prof.Dr., Pamukkale University
Other Study IDs: 13
Record Dates: First submitted 2023-06-30; First posted 2023-07-12 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Paraganglioma
Keywords: Paraganglioma; glomus
MeSH Terms: conditions — Paraganglioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine the head and neck paraganglioma cases treated in Pamukkale University hospital between 2007-2023 and improve our understanding of these cases and contribute to the knowledge surrounding head and neck paragangliomas.

DETAILED DESCRIPTION:
39 patients were selected and analyzed retrospectively. Demographic informations, complaints at the time of admission, radiological examinations, paraganglioma types, stages, postoperative complications, and relapsed cases were recorded.Preoperative staging plays a crucial role in surgical planning and predicting potential intraoperative complications. In such cases, combination therapy alongside surgery may improve treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of carotid paraganglioma
* Histopathological diagnosis of vagal paraganglioma
* Histopathological diagnosis of jugular paraganglioma
* Histopathological diagnosis of tympanic paraganglioma

Exclusion Criteria:

-Inadequate information in files

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent head and neck surgeries at Pamukkale University Hospital between 2007 and 2023, resulting in a histopathological diagnosis of paraganglioma
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Postoperative recurrence | may 2023-june 2023
  Incidence of recurrences after the surgery
Postoperative nerve paralysis | may 2023-june 2023
  Incidence of facial, vagus, hypoglossus, accesorius nerve paralysis after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No